CLINICAL TRIAL: NCT01601795
Title: Sevoflurane and Isoflurane - Cardioprotective Effects, Hemodynamic Stability and Pharmacokinetics During Cardiopulmonary Bypass With the MECC System
Brief Title: Sevoflurane and Isoflurane - During Cardiopulmonary Bypass With the MECC System (Minimized Extracorporeal Circuit)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University of Leipzig (Other); RWTH Aachen University (Other); Penn State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BS-57/12; Fassl_57/12 (Other: Universityhospital Basel_ANAESTHESIA_FASSL)
Record Dates: First submitted 2012-05-02; First posted 2012-05-18 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2014-01

CONDITIONS: Myocardial Reperfusion Injury
Keywords: Cardioprotection
MeSH Terms: conditions — Myocardial Reperfusion Injury | interventions — Sevoflurane; Isoflurane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sevoflurane (Active Comparator): During cardiopulmonary bypass, sevoflurane will be administered through a vaporizer integrated into heart-lung-machine.
  Interventions: Drug: Sevoflurane
- Isoflurane (Active Comparator): During cardiopulmonary bypass, isoflurane will be administered through a vaporizer integrated into heart-lung-machine.
  Interventions: Drug: Isoflurane

INTERVENTIONS:
Drug: Sevoflurane — volatile Anaesthetic, duration during cardiopulmonary bypass
  Other Names: Sevorane
  Arms: Sevoflurane
Drug: Isoflurane — volatile anesthetic, duration during cardiopulmonary bypass time
  Other Names: Isofluran
  Arms: Isoflurane

SUMMARY:
The use of volatile anesthetics in cardiac anesthesia is very common, because of their cardioprotective effects and their ability to ensure a sufficient depth of anesthesia. In line with the development of fast track concepts in cardiac anesthesia, volatile anesthetics are widely used to avoid a delayed recovery from cardiac surgery and anesthesia. Volatile anesthetics are delivered from calibrated vaporizers in the anesthesia machine or the cardiopulmonary bypass machine (during extracorporeal circulation).

Isoflurane and Sevoflurane are the most commonly used volatile anesthetics in patients undergoing cardiopulmonary bypass (CPB). The vaporizer of the anesthetics is on the cardiopulmonary bypass machine and the volatile agent is blended with air and oxygen. Until now, the pharmacokinetics of halothane, enflurane, isoflurane and desflurane during CPB have been described.

Sevoflurane might be of advantage because of additional myocardial protective effects during cardiac anesthesia and cardiopulmonary bypass. However, the pharmacokinetics of sevoflurane during CPB have not been investigated so far, although its being used at many hospitals.

The investigators will conduct a randomized prospective study with either sevoflurane or isoflurane during cardiopulmonary bypass surgery. The study will help to answer the questions about the possible cardioprotective effects of the widely used volatile anesthetics and the hemodynamic stability during cardiopulmonary bypass. Knowing the pharmacokinetics of these drugs allows the anesthesiologist to titrate the volatile anesthetics more precise.

The investigators hypothesizes that the maximal postoperative increase in troponin T will be smaller in the sevoflurane group than in the isoflurane group. The investigators hypothesizes that the total amount of noradrenaline needed during the entire period of cardiopulmonary bypass will be smaller in the sevoflurane group than in the isoflurane group. The investigators hypothesizes that kinetics of washin and washout at the CPB will be faster in the sevoflurane group than in the isoflurane group. The investigators hypothesizes that the time to extubation, respectively the length of stay in intensive care unit and hospital is shorter in the sevoflurane group than in the isoflurane group.

DETAILED DESCRIPTION:
Endpoints Primary Endpoint: Troponin

The study will compare the maximum postoperative troponin levels in the isoflurane and sevoflurane groups as a direct quantitative marker of damaged myocardial cells. Maximum troponin levels should be reached within the first 24 hours after surgery.

Secondary Endpoints:

A) Hemodynamic stability during on-pump

The investigators will compare the hemodynamic stability during CPB between the isoflurane and sevoflurane group. Therefore the total dosage of noradrenaline used during the surgery will be measured.

B) Washin and Washout Kinetic

Kinetics of washin and washout of sevoflurane and isoflurane during CPB will be investigated and described.

C) Extubation time and length of stay in the intensive care and in hospital

Time to extubation and the length of stay in intensive care unit and in hospital will be documented.

D) Mortality after 30 days

The mortality after 30 days will also be monitored. If the patient is no more in the hospital a phone call will be made.

ELIGIBILITY:
Inclusion Criteria:

* elective coronary bypass surgery
* preserved left ventricular function (LVEF (left ventricular ejection fraction) >55%)
* Age > 18 years
* planned MECC-System (minimized extracorporeal circulation)
* informed consent

Exclusion Criteria:

* chronic renal insufficiency (serum creatinine > 132umol/l)
* Body Mass Index > 35kg/m2
* additional operative procedures (eg. valve replacement/reconstruction)
* recent cardiac infarction (< 7 days) or elevated cardiac enzymes the day before surgery
* previous cardiac operation
* Pregnancy / Lactation
* known malignant hyperthermia (MH) or known relatives with MH
* known allergy against propofol, history of propofol infusion syndrome
* Drug abuse (cocaine, amphetamine, heroine, cannabis)
* non-judicious persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-07; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
postoperative maximum Troponin levels | 24 hours

SECONDARY OUTCOMES:
Hemodynamic stability during on-pump | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jens Fassl, MD, Principal Investigator — University Hospital Basel Departement of Anesthesiology and Intensive care medicine
Locations (1):
- University Hospital of Basel, Basel, Switzerland